CLINICAL TRIAL: NCT06056700
Title: Emotional Intelligence In Pregnancy and the Puerperium and Baby Blues Symptoms: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Norte (Other)
Collaborators: University of Wisconsin, Milwaukee (Other); University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13/2015
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Baby Blues Symptoms
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Women were informed of the study, and their participation was requested. Those who offered their willingness to participate signed the informed consent and were randomly assigned to the intervention group (IG) or the control group (CG). Randomization was performed using Microsoft Excel spreadsheet software. All study follow-up information was collected through this app. The information offered to all the mothers through the mobile application contained a welcome message, contact data, sociodemographic and clinical variables, and access to the TMM-24 questionnaire. However, the GI through the app had access to complementary information content regarding the CG. The mothers of the IG had additional training material related to the first two prenatal face-to-face training sessions and new information during the postnatal period throughout consecutive weeks 1 to 8.
  Interventions: Behavioral: Education
- Control Group (No Intervention): Women were informed of the study, and their participation was requested. Those who offered their willingness to participate signed the informed consent and were randomly assigned to the intervention group (IG) or the control group (CG). Randomization was performed using Microsoft Excel spreadsheet software. All study follow-up information was collected through this app. The information offered to all the mothers through the mobile application contained a welcome message, contact data, sociodemographic and clinical variables, and access to the TMM-24 questionnaire. However, the GI through the app had access to complementary information content regarding the CG. The mothers of the IG had additional training material related to the first two prenatal face-to-face training sessions and new information during the postnatal period throughout consecutive weeks 1 to 8.

INTERVENTIONS:
Behavioral: Education — All study follow-up information was collected through this app. The information offered to all the mothers through the mobile application contained a welcome message, contact data, sociodemographic and clinical variables, and access to the TMM-24 questionnaire. However, the GI through the app had access to complementary information content regarding the CG. The mothers of the IG had additional training material related to the first two prenatal face-to-face training sessions and new information during the postnatal period throughout consecutive weeks 1 to 8.
  Arms: Intervention Group

SUMMARY:
Background: Emotional intelligence pertains to the capacity for making decisions and adjusting to life's fluctuations, an attribute influenced by emotional conditions. Several scenarios impact nearly 80% of females, influencing their nurturing abilities. This study aimed to analyze the effectiveness of the "Happy in My Maternity" project in reducing baby blues symptoms in postnatal women. Methods: Employing a randomized clinical trial, hybrid interventions based on mobile application and i-person were conducted as part of an educational and emotional regulation curriculum. Enrollment encompassed the well-being of women. The program retained thirty-five participants, with thirty-four constituting the control cluster. The Trait-Meta Mood Scale (TMMS-24) questionnaire evaluation was administered to gauge emotional intelligence.

ELIGIBILITY:
Inclusion Criteria:

i) to have between 28 and 38 weeks of pregnancy, ii) pregnant women with follow-up and control at the participant hospital iii) women who signed their consent to participate in the study

Exclusion Criteria:

i) Women with high-risk pregnancies ii) Women suffering from psychiatric disorders before pregnancy such as anxiety, affective or disruptive behavior disorders

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Baby Blues Symptoms Relief | 14 weeks
  Baby Blues Symptoms Relief compared with the control group. These measurements were based on the Trait-Meta Mood Scale (TMMS-24) questionnaire evaluation for gauging emotional intelligence.

CONTACTS AND LOCATIONS:
Locations (1):
- Esmeralda Santacruz-Salas, Toledo, Castilla, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The IPD may be shared under anticipated requests.